CLINICAL TRIAL: NCT07152379
Title: An Open-label, Controlled Phase 2 Study Assessing a Challenge Transfusion of INTERCEPT Pathogen Reduced Red Blood Cells (RBCs) in Subjects With or Without Pre-existing Antibodies to INTERCEPT RBCs
Brief Title: Challenge Transfusion of INTERCEPT Pathogen Reduced Red Blood Cells (RBCs) in Subjects With or Without Pre-existing Antibodies to INTERCEPT RBCs
Acronym: Challenge
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cerus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CLI 00177
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Transfusion Reaction, Hemolytic
Keywords: INTERCEPT, red blood cells, antibody
MeSH Terms: conditions — Transfusion Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Subjects with Antibodies to INTERCEPT RBC Either Naturally Acquired or Treatment Emergent (Experimental): Test subjects will be selected from the pool of subjects who have documented antibodies to INTERCEPT RBC either naturally acquired (e.g., detected during a pre-transfusion enrollment screening process) or treatment-emergent following an INTERCEPT RBC transfusion. Eligible subjects may have been enrolled in either the Test or Control arms of prior studies; subjects whose randomization status is still blinded may also be enrolled in this study if they have completed the study requirements of the prior study and >120 days have elapsed since exposure to a study RBC product.
  Interventions: Device: INTERCEPT RBCs
- Subjects with history of transfusion without INTERCEPT RBC antibodies (Active Comparator): Control subjects will be identified by participating study sites as individuals with a history of allogeneic transfusion(s) without a history of or currently demonstrable INTERCEPT RBC antibodies.
  Interventions: Device: INTERCEPT RBCs

INTERVENTIONS:
Device: INTERCEPT RBCs — Transfusion of fresh (≤14 days old) allogeneic INTERCEPT RBCs.

SUMMARY:
This study aims to determine whether transfusion of INTERCEPT RBCs into patients with pre-existing antibodies to INTERCEPT RBCs will result in increased antibody titer indicative of a secondary immune response, and whether these immune responses would be associated with clinical adverse events, increased RBC clearance, and/or evidence of hemolysis. Because the recovery and survival of fresh allogeneic INTERCEPT RBCs in patients with a diverse group of diseases is poorly characterized, a Control group of subjects without a history or evidence of antibodies to INTERCEPT RBCs may be evaluated as a comparator (Control group subjects may or may not have previously been transfused with INTERCEPT RBCs).

The study will also compare and correlate results from anti-human globulin (AHG) crossmatch using INTERCEPT RBCs prepared for transfusion, with results from indirect antiglobulin testing (IAT) with S 303 treated reagent RBCs (i.e., INTERCEPT RBC screening assay, as used in previous studies) to assess the utility of the AHG crossmatch to define the compatibility of transfused INTERCEPT RBCs

DETAILED DESCRIPTION:
This is a prospective, open-label, controlled Phase 2 study. Consented subjects will be screened for currently detectable or previously documented allogeneic, autologous, and INTERCEPT RBC-specific antibodies, assigned to a study arm, then receive a small volume transfusion of fresh (≤14 days old) allogeneic INTERCEPT RBCs under careful clinical oversight for adverse events including evidence of hemolysis.

Subjects will have blood samples drawn pre-transfusion and over 90 days after transfusion (Days 0, 1, 7, 14, 30, 60, and 90) to detect evidence of primary or secondary immune responses to INTERCEPT RBCs (see Section 8.4.2), and to assess the in vivo post transfusion 24-hour recovery (PTR24) and survival assessed as the half-life [T50], predicted mean/median lifespan, and area-under-the-survival curve (AUC) of the transfused cells.

RBCs and plasma will be collected and stored frozen for further analysis. Specific studies will include gel card-based INTERCEPT RBC antibody screen assay and titer, AHG crossmatch using cells from INTERCEPT RBC units prepared for transfusion, as well as RBC flow cytometric analysis using an antibody specific for acridine to quantitate the proportion of circulating INTERCEPT RBCs and the acridine adduct surface density.

Clinical evidence of hemolysis will be evaluated using routine laboratory tests, including complete blood counts (CBC), chemistry tests and urinalysis.

Test and Control subjects may be recruited from other INTERCEPT RBC studies. Control subjects may be recruited from specific age groups (e.g., children, adults) with specific medical conditions that are known to impact RBC survival in vivo, particularly conditions that are shown to be present in Test subjects (e.g., sickle cell disease, thalassemia).

After an initial challenge dose of 30-40 ml total volume (appx 20 ml RBCs at 50-70% hematocrit), subjects may be consented and enrolled for second and third challenge doses after completion of all study requirements for the subject's prior dose as well as a 120-day minimum wash-out period since the previous study transfusion.

If a subject requires a therapeutic RBC transfusion, had no evidence of hemolysis with the previous challenge dose(s) and remains eligible for a subsequent challenge dose, they may be administered a challenge dose of one full unit volume. Prior to administering each full unit challenge dose, a Data Safety Monitoring Board (DSMB) must perform an interim safety analysis considering all available study data.

Subjects may receive up to three challenge doses of INTERCEPT RBCs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥4 years in children who meet the requirement of US Code of Federal Regulation (CFR) Title 21, §50.53 as determined by the local Institutional Review Board (IRB).
* Control subjects shall have no current or previously documented antibodies to INTERCEPT RBC.
* Test subjects shall have current or previously documented natural or treatment-emergent antibodies to INTERCEPT RBCs.
* History of prior transfusion with allogeneic blood products (INTERCEPT or non-INTERCEPT treated).
* >120 days from the subjects most recent exposure to Study RBCs (pathogen reduced or non-pathogen reduced - if any) prior to the planned study transfusion.
* Signed and dated informed consent form

Exclusion Criteria:

* Foreseeable active blood loss due to trauma, surgery, or pathologic condition during the study period.
* Exposure to another interventional drug or device in a clinical study within 28 days prior to enrollment or concurrently during the study.
* Positive Direct Antiglobulin Test (≥2+) at the time of screening, prior to the first study transfusion.
* Current or historical medical conditions judged by the Investigator to significantly increase the risk of morbidity/mortality due to hemolysis or the medical management of acute hemolysis.
* Treatment with any medication known to affect RBC viability at the time of enrollment (e.g., ribavirin, sulfa drugs, chemotherapy medications, methylene blue, dapsone, levodopa, methyldopa, nitrofurantoin and its derivatives, phenazopyridine, quinidine, and hydantoins)
* History of or development of a drug-associated RBC antibody not associated with INTERCEPT RBCs.
* Congenital or acquired immunodeficiency judged by the Investigator to potentially impact the humoral immune response.
* Immunosuppressive therapy within 1 month prior to enrollment or during the study period, including steroids and intravenous immunoglobulin.
* Current or historical RBC alloantibodies that are judged by the Investigator to prevent selection of antigen-negative RBCs for transfusion.
* History of immunoglobulin A (IgA) deficiency, severe allergic reaction to blood product(s), or clinical requirement to receive washed cellular products.
* History of warm autoantibody with hemolysis.
* Subjects who are pregnant, or biologically able to become pregnant and unwilling to remain on medically accepted contraception during this study.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Acute or delayed hemolytic transfusion reactions | 90 days
  Incidence of acute or delayed hemolytic transfusion reactions (AHTR or DHTR) attributed to the study INTERCEPT RBC transfusion, based upon clinical and/or laboratory findings, using Centers for Disease Control (CDC) Hemovigilance criteria.
Clearance | 30 days
  Incidence of rapid clearance (complete clearance by Day 30) of INTERCEPT RBCs assessed by flow cytometry.

SECONDARY OUTCOMES:
Increase in Antibody Titer | 90 days
  Incidence of ≥4-fold increase in titer of INTERCEPT RBC antibodies from baseline (≥2 doubling dilution increase in titer), indicative of a secondary immune response.
In vivo recovery and survival kinetics | 90 days
  In vivo recovery and survival kinetics of INTERCEPT RBCs (PTR24, lifespan, T50 and AUC) in the presence and absence of INTERCEPT RBC antibodies.
  In vivo recovery and survival kinetics of INTERCEPT RBCs (PTR24, lifespan, T50 and AUC) in the presence and absence of INTERCEPT RBC antibodies.
Immunoglobulin subclass of INTERCEPT RBC-bound antibodies | 90 days
  Presence of and immunoglobulin subclass of INTERCEPT RBC-bound antibodies assessed by flow cytometry.
RBC alloantibodies or autoantibodies | 90 Days
  RBC alloantibodies or autoantibodies not specific to INTERCEPT RBCs that develop during the study period.
Antibody Characterization | 90 Days
  Characterization of INTERCEPT RBC antibodies before and after challenge transfusion including: titer, binding specificity, immunoglobulin class, immunoglobulin subtype, and monocyte monolayer assay test result.
Characterization of membrane-bound acridine | 90 Days
  Characterization of membrane-bound acridine (acridine molecules per RBC) over the lifespan of transfused INTERCEPT RBCs in the presence and absence of INTERCEPT RBC antibodies.
Comparison of AHG Crossmatch and INTERCEPT RBC antibody indirect antiglobulin test | Day 0
  Percent positive/negative agreement between pre-transfusion AHG crossmatch and INTERCEPT RBC antibody indirect antiglobulin test results with undiluted as well as serially diluted subject plasma.

OTHER OUTCOMES:
Proportion of subjects with Adverse Events (AEs) | 24 hours after transfusion
  Proportion of subjects with AEs (non-serious and serious) documented from the start of the study RBC transfusion up to 24 hours after transfusion of any INTERCEPT RBC challenge.
Proportion of subjects with related AEs | 90 Days
  Proportion of subjects with possibly, probably, or definitely related adverse events (i.e., transfusion reactions [TR]) documented from the start of the study RBC transfusion until the end of Day 90 (+/- 7 days).
Proportion of subjects with study transfusion related serious adverse events (SAEs) | 90 Days
  Proportion of subjects with study transfusion possibly, probably, or definitely related SAEs documented from the start of the study RBC transfusion until the end of the 90-day (+/- 7 days) post-transfusion monitoring period.